CLINICAL TRIAL: NCT03623178
Title: Assertive Community Treatment for Patients Suffering From Substance Use
Brief Title: Assertive Community Treatment for Patients Suffering From Substance Use Disorders
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Louise Penzenstadler, Principal investigator, University Hospital, Geneva
Other Study IDs: ID 2017-01087
Record Dates: First submitted 2018-08-01; First posted 2018-08-09 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2018-08

CONDITIONS: Substance Use Disorders
Keywords: Substance Use Disorders; Assertive Community Treatment; Community Treatment; Treatment engagement; Service Use
MeSH Terms: conditions — Substance-Related Disorders | interventions — Community Mental Health Services

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Assertive Community Treatment: patients with DSM-5 Diagnosis of SUD and one of the following criteria (1) present important functional difficulties, in at least one of the following areas: everyday life activities and maintaining a supportive social network, for minimum two years.
  or (2) difficulties to attend their health care appointments, during the last 3 months.
  Interventions: Other: Assertive Community Treatment

INTERVENTIONS:
Other: Assertive Community Treatment — The intervention program is a type of very flexible community treatment. This is facilitated by a small case load ratio per health care professional (1:10). The healthcare workers are specialized in SUD treatment. The time of the intervention differs, there is no prefixed limitation but the duration of the intervention depends on the goals agreed on with the patient. The main objective of this intervention is to ensure an adherence to an addiction treatment program and establish or consolidate a stable healthcare and social network for the patient. The intervention aims to prevent service disengagement. The healthcare workers will explore specific patient needs and ensure that health and social services are better coordinated to fit their needs.

SUMMARY:
According to the World Health Organization the population suffering from addiction problems is increasing. This population is characterized by multiple needs at the medico-psychosocial level. However, some of these patients, a particular subgroup that we are going to be interested in the so-called "high need" user group, find it difficult to access and stay in outpatient treatment programs. Persons with substance use disorder often present a chaotic use of the health system, including a high number of hospitalizations in times of crisis. These individuals also show very low utilization of health care services, accompanied by social marginalization. This can be related to relapses and poor social functioning. A high number of relapses occur particularly at the end of hospitalization. Community Interventions, such as Assertive Community Treatment (ACT) should increase the adherence of these patients to treatment by accompanying them in the community and helping them during sensitive and crisis periods. One of the objectives of the study is to evaluate the impact of ACT on the time until service disengagement, measuring treatment adherence. The secondary objectives of this study will be to see the effect of ACT on duration and type of hospitalizations, as well as the number of emergency room visits. The investigators will focus on the impact of ACT on the participant's medico-psycho-social network, substance use and other psychological variables. The investigators will also evaluate his or her psychiatric symptoms and global and social functioning. Life satisfaction and satisfaction with the care received will also be measured. The study will investigate this through questionnaires at the beginning of care, at three months, six months and 12 months after the start of the ACT intervention.

ELIGIBILITY:
Inclusion Criteria:

* Substance use disorder
* Competent subjects, able to give informed consent
* French speaking

Exclusion Criteria:

* Evidence of organic brain disease or learning disability based on the chart review.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subgroup of high need users with difficulties in engaging in substance use disorder treatment.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Treatment adherence | at 12 months
  Number of days until service disengagement

SECONDARY OUTCOMES:
Service use | at 12 months
  Number of hospital admissions and number of days in hospital
Patient network | 0, 3, 6, 12 months
  Number of persons in network
Number of ER visits | 0, 3, 6, 12 months
  Number of ER visits reviewed on patient file
Addictive behaviour | 0, 3, 6, 12 months
  Alcohol, Smoking and Substance Involvement Screening Test (ASSIST. V.3 French)
General psychiatric symptoms | 0, 3, 6, 12 months
  Health of Nation Outcome Scale - French version (HoNOS-F): scores 0 - 52 (higher score = more psychiatric symptoms)
Global Functioning | 0, 3, 6, 12 months
  World Health Organization Disability Assessment Schedule (WHODAS)
General life satisfaction: Satisfaction With Life Scale | 0, 3, 6, 12 months
  Satisfaction With Life Scale: scores 5 - 35 (higher score = higher life satisfaction)

OTHER OUTCOMES:
Patient satisfaction with Assertive Community Treatment | at 3, 6, 12 months
  Patient satisfaction with Assertive Community Treatment (very satisfied, satisfied, more or less satisfied, not satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Louise Penzenstadler, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Service d'addictologie, HUG, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No